CLINICAL TRIAL: NCT00454233
Title: A Randomized, Double Blind, Placebo and Active Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability and Potential Efficacy of a 12-Week Treatment With YM543 in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Safety and Efficacy Study With YM543 in Type 2 Diabetes Mellitus Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 543-CL-003; EudraCT number: 2006-001110-33
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2; YM543; Treatment; Safety; efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): Dose 1
  Interventions: Drug: YM543
- 2 (Experimental): Dose 2
  Interventions: Drug: YM543
- 3 (Experimental): Dose 3
  Interventions: Drug: YM543
- 4 (Experimental): Dose 4
  Interventions: Drug: YM543
- 5 (Active Comparator)
  Interventions: Drug: Metformin
- 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM543 — Oral
  Arms: 1; 2; 3; 4
Drug: Metformin — Oral
  Arms: 5
Drug: Placebo — oral
  Arms: 6

SUMMARY:
The purpose of this study is to investigate the safety of YM543 in type 2 Diabetes Mellitus patients and to investigate whether this study drug is effective in these patients

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive subjects diagnosed with T2DM
* Stable diet and exercise program for at least 6 weeks
* Inadequate glycemic control indicated by HbA1c and FPG level at Visit 1

Exclusion Criteria:

* Any known complication of T2DM indicating a late disease state, clinical manifestations of macro- and/or micro vascular disorders
* Use of insulin or oral blood glucose lowering drugs in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (adverse events; biochemical, hematological and urine analysis tests; vital signs, 12-lead ECG, physical examination) | 3 Months

SECONDARY OUTCOMES:
Efficacy and pharmacodynamics (change in HbA1c and fasting plasma glucose; change in urinary glucose excretion; plasma levels of YM543; C-peptide, insulin, fructosamine, non-esterified fatty acids, triglyceride, cholesterol-panel) | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (6):
- Russia (6):
  - 4 Sites, Moscow
  - Nizhny Novgorod
  - Petrozavodsk
  - 10 Sites, Saint Petersburg
  - Samara
  - Yekaterinburg